CLINICAL TRIAL: NCT04054531
Title: An Open-label, Phase II Study of KN046 Evaluating the Efficacy and Safety of KN046 Plus Platinum-based Doublet Chemotherapy as First Line Therapy in Advanced Non-small Cell Lung Cancer Subjects.
Brief Title: Study of KN046 With Chemotherapy in First Line Advanced NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KN046-202
Record Dates: First submitted 2019-08-06; First posted 2019-08-13 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-08

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KN046 + carboplatin/paclitaxel (Experimental): KN046 5 mg/kg IV every three weeks (Q3W) +Carboplatin AUC5 IV Q3W x 4 cycles + Paclitaxel 500 mg/m2 IV Q3W x 4 cycles
  Interventions: Biological: KN046; Drug: Paclitaxel; Drug: Carboplatin
- KN046 + carboplatin/pemetrexed (Experimental): KN046 5 mg/kg IV Q3W +Carboplatin AUC5 IV Q3W x 4 cycles + Pemetrexed 500 mg/m2 IV Q3W x 4 cycles
  Interventions: Biological: KN046; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Biological: KN046 — IV infusion
Drug: Paclitaxel — IV infusion
  Arms: KN046 + carboplatin/paclitaxel
Drug: Pemetrexed — IV infusion
  Arms: KN046 + carboplatin/pemetrexed
Drug: Carboplatin — IV infusion

SUMMARY:
This is a phase II study of KN046 plus platinum-based doublet chemotherapy in previously untreated advanced non-squamous and squamous NSCLC subjects.

The study will assess primarily the safety and efficacy of KN046 plus platinum-based doublet chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of stage IV NSCLC;
* Has not received prior systemic treatment for metastatic NSCLC;
* Has measurable disease based on RECIST 1.1.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* Has adequate organ function.
* Has provided tumor tissue from locations not radiated prior to biopsy.

Key Exclusion Criteria:

* Previous immunotherapy (e.g. anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways)
* Previously untreated or symptomatic central nervous system (CNS) metastases
* Has received a live-virus vaccination within 28 days of planned treatment start.
* Previously had a severe hypersensitivity reaction to treatment with another monoclonal antibody and chemotherapy.
* Has or had active autoimmune disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 12 months
  ORR was defined as the percentage of participants who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) as assessed by RECIST 1.1. ORR.
Duration of Response (DOR) as Assessed by Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) | Up to approximately 12 months
  For participants who demonstrated a confirmed response (Complete Response [CR]: Disappearance of all target lesions or Partial Response [PR]: At least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of CR or PR until disease progression as assessed by RECIST 1.1 or death.

SECONDARY OUTCOMES:
Number of Participants Who Experienced a treatment-emergent adverse event (TEAE) | Up to approximately 12 months
  TEAE was defined any treatment emergent adverse event.
Number of Participants Who Experienced an immune-related AE (irAE) | Up to approximately 12 months
  irAE was defined any immune-related adverse event (AE).

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhao Y, Chen G, Li X, Wu J, Chang B, Hu S, Yang S, Xu T, Liu Y, Wang N, Zhang L, Huang Y. KN046, a bispecific antibody against PD-L1 and CTLA-4, plus chemotherapy as first-line treatment for metastatic NSCLC: A multicenter phase 2 trial. Cell Rep Med. 2024 Mar 19;5(3):101470. doi: 10.1016/j.xcrm.2024.101470. PMID 38508135